CLINICAL TRIAL: NCT03187912
Title: Effect-evaluation of an Accelerated Corneal Cross-linking Protocol With Different Riboflavin Solutions
Brief Title: Accelerated Corneal Cross-linking With Different Riboflavin Solutions
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Gerald Schmidinger, Ass. Prof. PDDr., Medical University of Vienna
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 1390/2016
Record Dates: First submitted 2017-06-12; First posted 2017-06-15 (Actual); Last update posted 2021-03-03 (Actual); Status verified 2021-03

CONDITIONS: Keratoconus
MeSH Terms: conditions — Keratoconus | interventions — Riboflavin

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Riboflavin with 20% Dextran (Active Comparator): Riboflavin drops with Dextran
  Interventions: Drug: Riboflavin
- Riboflavin with HPMC (Active Comparator): Riboflavin drops with HPMC
  Interventions: Drug: Riboflavin

INTERVENTIONS:
Drug: Riboflavin — Riboflavin with 20% Dextran or HPMC will be admininstered every 2 minutes for overall 30 minuts (Dextran) or 10 minutes (HPMC), respectively

SUMMARY:
Following the Bunsen-Roscoe law, accelerated cross-linking protocols with higher irradiation intensities and shorter irradiation times have been introduced. In addition, new riboflavin solutions with HPMC (hydroxylpropyl methylcellulose) instead of dextran found its way into CXL-treatment. The aim of this trial is to evaluate clinical outcomes in an accelerated corneal collagen cross-linking protocol with different riboflavin solutions.

ELIGIBILITY:
Inclusion Criteria:

* Progressive Keratoconus
* Indication for treatment
* Preoperative Pachymetry > 400

Exclusion Criteria:

* Pregnancy
* Re-CXL
* Keratitis
* Other visual acuity limiting eye diseases than corneal ectatic diseases

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2016-09-19 (Actual); Primary Completion 2020-03-30 (Actual); Study Completion 2020-03-30 (Actual)

PRIMARY OUTCOMES:
Kmax | 12 months
  Steepest Keratometry

SECONDARY OUTCOMES:
Postoperative central stromal depth of the Demarcation Line | 1 month
  The depth of the Demarcation Line after CXL will be measured one month postoperatively with an AS-OCT
LogMAR | 12 months
  Visual Acuity

CONTACTS AND LOCATIONS:
Locations (1):
- Medical University of Vienna, Department of Ophthalmology, Vienna, Austria